CLINICAL TRIAL: NCT01381419
Title: A Single-blind, Randomised, Placebo-controlled, Ascending Dose Study to Evaluate the Safety, Tolerability and Pharmacokinetics of GSK1144814 in Healthy Male and Female Subjects and an Open-label Positron Emission Tomography Study in Healthy Male Subjects to Evaluate the Neurokinin-1 (NK1) Receptor Occupancy of GSK1144814 in the Living Human Brain Using 11C GR205171.
Brief Title: First Time in Human Study (FTIH) With Positron Emission Tomography (PET)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 111321
Record Dates: First submitted 2011-06-09; First posted 2011-06-27 (Estimated); Last update posted 2017-07-07 (Actual); Status verified 2017-07

CONDITIONS: Schizophrenia
Keywords: pharmacokinetics; safety; positron emission tomography (PET); single ascending dose
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Part A, Cohort 1 (Experimental): In Cohort 1, four subjects (two on active and two on placebo for first dose, and then three on active and one on placebo for subsequent doses) will be included. Subjects will be dosed at least 30 minutes apart over the dosing day and only doses administered where the predicted plasma concentration will remain below those corresponding to the MABEL.
  Interventions: Drug: GSK1144814
- Part A, cohort 2 (Experimental): In Cohort 2, 10 subjects will be included (8 active : 2 placebo). Dosing will start once the previous cohort (Cohort 1) has completed the Treatment Phase. For Cohort 2 and any subsequent cohorts, dosing will take place on two different days when a new dose is administered such that no more than one subject receives the agreed ascending dose on the first dosing day. Doses may be split in up to three divided doses given 2 to 3 hours apart. Dosing for the first four sessions in each cohort will be staggered over 2 days. On the first day of each dosing session, only one subject will receive the highest dose for that dosing session and at least one subject each will receive placebo. The remaining subjects in the cohort will be dosed on the second day according to the randomisation plan.
  Interventions: Drug: GSK1144814
- Part B (Experimental): Part B of the study will consist of a Screening Visit (up to 30 days before the dosing session), three PET scans (where possible, all three scans may be performed in one visit when subject is admitted overnight) and a Follow-up Visit. Each subject will receive an oral dose of study drug. The dose may be split in up to three divided doses given 2 to 3 hours apart.
  Interventions: Drug: GSK1144814

INTERVENTIONS:
Drug: GSK1144814 — Single dose.
  Arms: Part A, Cohort 1
Drug: GSK1144814 — Single dose which may be split in up to three divided doses given 2 to 3 hours apart.
  Arms: Part A, cohort 2
Drug: GSK1144814 — Single dose that may be split in up to three divided doses given 2 to 3 hours apart.
  Arms: Part B

SUMMARY:
This study described in the present protocol consists of two sections. Part A is the first administration into man to evaluate the safety, tolerability and pharmacokinetics of single ascending doses of GSK1144814. The study is a single-blind, randomised, placebo-controlled design in healthy male and female (of non-childbearing potential) subjects. Part B will be an open-label design in healthy male subjects to assess the GSK1144814 neurokinin-1 (NK1) receptor occupancy by positron emission tomography (PET) scanning with [11C]-GR205171

DETAILED DESCRIPTION:
GSK1144814 is a dual neurokinin-1 (NK1) and neurokinin-3 (NK3) antagonist with the potential to treat schizophrenia & depression.

This study described in the present protocol consists of two sections. Part A is the first administration into man to evaluate the safety, tolerability and pharmacokinetics of single ascending doses of GSK1144814. The study is a single-blind, randomised, placebo-controlled design in healthy male and female (of non-childbearing potential) subjects. Part B will be an open-label design in healthy male subjects to assess the GSK1144814 NK1 receptor occupancy by positron emission tomography (PET) scanning with [11C]-GR205171.

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by a responsible physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if, in the opinion of the Investigator, the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Male or female aged between 18 and 55 years (inclusive) for Part A, or male aged between 25 and 55 years (inclusive) for Part B.
* A female subject is eligible to participate in Part A if she is of:

  • Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea (in questionable cases a blood sample with simultaneous follicle stimulating hormone [FSH] >40 mIU/mL and oestradiol <40 pg/mL [<140 pmol/L] is confirmatory). Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to discontinue HRT to allow confirmation of post-menopausal status prior to study enrolment. For most forms of HRT, at least 2 to 4 weeks will elapse between the cessation of therapy and the blood sampling; this interval depends on the type and dosage of HRT. Following confirmation of their post-menopausal status, they can resume the use of HRT during the study without the use of a contraceptive method.
* A male subject must agree to use one of the contraception methods listed in Section 8.1. This criterion must be followed from the first investigational product dosing day until at least 3 months after receiving the last dose of the investigational product.
* Body weight ≥50 kg and body mass index (BMI) within the range 18 to 29.9 kg/m2 (inclusive).
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* QTcB or QTcF <450 msec.
* Demonstrates no evidence of mental impairment or co-morbid psychiatric disorders.

Exclusion Criteria:

* The subject has a positive pre-study drug/alcohol screen. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates, cannabinoids and benzodiazepines.
* A positive pre-study hepatitis B surface antigen (HBsAg) or positive hepatitis C virus (HCV) antibody test result within 3 months of Screening.
* A positive test result for antibodies to human immunodeficiency virus (HIV)-1/2.
* Significant renal abnormality (from medical history or as indicated by laboratory investigations. In addition, subjects with idiopathic haematuria or proteinuria or conditions such as benign orthostatic proteinuria and benign familial haematuria should be excluded from the study).
* History of regular alcohol consumption within 6 months of the study start defined as:

  • An average weekly intake of greater than 21 units or an average daily intake of greater than 3 units (males), or defined as an average weekly intake of greater than 14 units or an average daily intake of greater than 2 units (females). One unit is equivalent to a half-pint (220 mL) of beer or 1 measure (25 mL) of spirits or 1 glass (125 mL) of wine.
* The subject has participated in a clinical trial and has received an investigational product within 3 month prior to the first investigational product dosing day in the current study.
* Exposure to more than four new chemical entities within 12 months prior to the first investigational product dosing day.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to receiving the first dose of the investigational product, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* History of sensitivity to any of the investigational products, or components thereof or a history of drug or other allergy that, in the opinion of the Investigator or GSK Medical Monitor, contraindicates their participation in the study.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56-day period.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* History or presence of clinically significant cardiac arrhythmias, or other clinically significant cardiac disease.
* Smokers confirmed by a positive urinary cotinine test (greater than the local laboratory lower limit of quantification [LLQ] of 200 ng/mL or lower). Urine cotinine levels will be measured during Screening and at Baseline.
* Consumption of Seville oranges (including marmalade) and/or grapefruit and/or Chinese grapefruit (pomelo) and/or grapefruit hybrids and/or exotic citrus fruits and/or their fruit juices from 7 days prior to the first investigational product dosing day.
* Consumption of red wine from 7 days prior to the first investigational product dosing day

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2008-10-20 (Actual); Primary Completion 2009-04-01 (Actual); Study Completion 2009-04-01 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability: Adverse event monitoring, vital signs (blood pressure, heart rate, respiratory rate, oral body temperature, ECGs (12 lead and Holter), clinical laboratory assessments (standard laboratory parameters). | 2 months
Pharmacokinetics: time-point immediately prior to the first quantifiable plasma concentration (tlag), Cmax, time of occurrence of Cmax (tmax), AUC from time zero (pre dose) to the time of the last quantifiable concentration (AUC0-infinity), | 72 hours
Volume of distribution (VT) of [11C] GR205171 in the brain at Baseline and following oral doses of GSK1144814. | 7 days
NK1 receptor occupancy in the brain at Baseline and following oral doses of GSK1144814. | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Harrow, Middlesex, United Kingdom

REFERENCES:
- See also: Results for study 111321 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/111321?search=study&study_ids=111321#rs